CLINICAL TRIAL: NCT01767597
Title: Is the Combination of Screening Algorithms and Use of Hepatitis B Rapid Tests Useful in Optimizing the Screening and Prevention of Hepatitis B?
Brief Title: Application of HBV Rapid Tests as a Tool for Wide-Use Screening
Acronym: OPTISCREEN-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Gilead Sciences (Industry); Roche Pharma AG (Industry); Mairie de Paris (Unknown); BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IMEA 38; 2011-A01603-38 (Registry Identifier: ANSM)
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis B; Liver Cirrhosis; Carcinoma, Hepatocellular
Keywords: rapid test; screening; ELISA; hepatitis B virus; access to care
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELISA testing (Active Comparator): HBV infection status determined by enzyme-linked immuno-assay (ELISA)
  Interventions: Other: ELISA testing
- Rapid testing (Experimental): HBV infection status determined initially by a rapid test, then confirmed by enzyme-linked immuno-assay (ELISA).
  Interventions: Other: ELISA testing; Other: Rapid testing

INTERVENTIONS:
Other: ELISA testing — Enzyme-linked immuno-assay (ELISA) will be used to determine hepatitis B surface antigen (HBsAg) and anti-HBsAg antibody (anti-HBs Ab) status. Results will be given after test results are available (8-10 days).
Other: Rapid testing — A rapid test will be performed to determine the subjects' hepatitis B surface antigen (HBsAg, using VIKIA®) and anti-HBs antibody status (anti-HBs Ab, using Quick ProfileTM). Results will be given the same day.
  Other Names: VIKIA®, Biomerieux, Marcy-l'Étoile, France; Quick ProfileTM, Lumiquick, Santa Clara, CA, USA
  Arms: Rapid testing

SUMMARY:
With over 280 000 chronic carriers, 2,500 new annual cases and 1,300 deaths each year, hepatitis B is currently a frequent and potentially severe disease in France, despite efforts towards prevention and effective care.

In terms of prevention, France has very low immunization coverage (27.7%) and a high percentage of people ignoring HBV status (55%), leading to a delay in care. This is partly explained by poor knowledge of hepatitis B infection in the general population and an underestimation of the health impact of hepatitis B by doctors and health officials. Until recently, there have been no national guidelines governing its implementation (which is variable depending on the structures where screening is performed) and an insufficient evaluation of screening practices. Thus, data on the severity of liver disease, indications for treatment of HBV-infected patients and data on the use of vaccination for nonimmunized people are scarce. Furthermore, while HIV rapid tests are beginning to be used more widely, particularly to address the issue of people who do not come back and collect their results and to better adapt "counselling", their usefulness to detect of hepatitis B virus has not been evaluated to date.

The main objective of the Optiscreen B Study is to determine the benefit, if any, of using rapid tests as a screening tool to improve diagnosis, care and prevention of hepatitis B. Individuals risk of HBV-infection will be randomized into 2 groups, one group for which screening will be performed by usual serological test and a second group for which screening will be based on rapid tests. Centers will be selected to represent a diverse range of health centers whose aims include screening, prevention and/or vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Born in a country of middle or high HBV endemicity
* Parents born in a country of middle or high HBV endemicity
* Travellers or residents from a country of middle or high HBV endemicity
* Blood, organ, tissue, sperm, and/or ovary donners or candidate donners.
* Health-care workers suspected of coming into direct contact with an HBV-infected individual and/or exposed to blood or any biological products from an HBV-infected individual
* Close contact with HBsAg-positive individuals (living in the same household, sexual partner, sharing needles, etc.)
* Individuals with accidental exposure to HBV
* Individuals with multiple sexual partners
* Men who have sex with men
* Pregnant women
* Hemodialysis
* Individuals requiring immunosuppressive therapy
* Individuals with persistently elevated transaminase levels
* HIV-positive
* Intravenous drug users

Exclusion Criteria:

* Age <18 years old
* Not capable of providing informed consent
* Already participated in a multi-center validation of HBV rapid tests
* Having, in their possession, irrefutable results of a prior test for hepatitis B virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bottero, MD, Principal Investigator — Hôpital Saint-Antoine
Locations (5):
- France (5):
  - Centre de Santé au Maire-Volta, Paris
  - Centre d'examen de santé de la CPAM, antenne rue du Maroc, Paris
  - Consultation Policlinique de l'hôpital Saint-Antoine, Paris
  - Consultation Voyage de l'hôpital Saint-Antoine, Paris
  - CDAG de Belleville, Paris

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon official request by interested parties. All requests are subject to approval by the Scientific Committee.

REFERENCES:
- [Result] Bottero J, Boyd A, Gozlan J, Carrat F, Lemoine M, Rougier H, Varsat B, Boo N, Charlois-Ou C, Collignon A, Cha O, Campa P, Dhotte P, Girard PM, Lacombe K. Effectiveness of hepatitis B rapid tests toward linkage-to-care: results of a randomized, multicenter study. Eur J Gastroenterol Hepatol. 2016 Jun;28(6):633-9. doi: 10.1097/MEG.0000000000000620. PMID 26954517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 29 February 2012 to 5 July 2012, volunteers were recruited from five study centers in the Paris metropolitan region, which actively participate in HBV screening, vaccination, and care - two sexually transmitted disease clinics, one primary healthcare center, one general screening center, and one travel clinic.
Pre-assignment Details: 2061 participants were initially screened for eligibility. Of them, 625 did not meet inclusion criteria and 436 declined to participate. In total, 1000 participants were randomized.
Period: Overall Study
Arm/Group | ELISA Testing | Rapid Testing
Started | 500 | 500
Completed | 496 | 499
Not Completed | 4 | 1
Not completed — Incomplete intervention | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants completing their intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | ELISA Testing | Rapid Testing | Total
Number analyzed (Participants) | 496 | 499 | 995
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (16.0) | 40.1 (15.6) | 40.4 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 272 | 522
  Male | 246 | 227 | 473
HBV prevalence of birth country [Number; unit: participants]
  Low (<2.0%) | 292 | 275 | 567
  Intermediate (2.0-8.0%) | 116 | 137 | 253
  High (>8.0%) | 88 | 87 | 175
Health insurance plan [Number; unit: participants]
  Social security | 465 | 472 | 937
  CMU | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Appropriately Seeking Care
Description: Subjects who are considered required to seek further care are as follows:
  * those who need HBV vaccination (non-immunized)
  * those who are infected with hepatitis B virus (infected)
  Of these patients, subjects who have achieved appropriate care are considered as follows:
  * non immunized subjects who have initiated HBV vaccination sequence (vaccinated)
  * infected subjects who seek health care at a specialized center, allowing to quantify the severity of liver-related disease (infected with care)
  The percentage of patients appropriately seeking care will be then calculated by the following formula:
  ((nb Vaccinated + nb infected with care) / (nb non-immunized + nb infected))*100
Time Frame: 6 months
Population: Only participants needing further medical intervention were included in analysis: non-immunized (HBsAg negative, anti-HBc antibody negative, anti-HBs antibody negative) or infected (HBsAg positive).
Measure: Number; unit: percentage of participants
Arm/Group | ELISA Testing | Rapid Testing
Number analyzed (Participants) | 211 | 198
percentage of participants | 5.7 | 4.0
Statistical Analysis 1: Comparison: ELISA Testing vs Rapid Testing; Power calculations were performed to detect >15% difference in immediate linkage-to-care and vaccination. We hypothesized from discussions with an expert panel that ~30% of participants would have appropriate care with standard HBV serology. Assuming type 1 error=0.05 and power=80%, 152 participants per arm would be needed. As ~40% of the population would be nonimmunized or HBsAg-positive from previous data, a minimum 375 participants per arm would be required; Test type: Superiority or Other; p = 0.5, Chi-squared — No p-value adjustments for multiple comparisons were required. Significance was determined using a p-value <0.05

ADVERSE EVENTS:
Time Frame: 6 months
Description: Any event possibly related to physical HBV test.
Arm/Group | ELISA Testing | Rapid Testing
Serious Adverse Events (participants affected / at risk) | 0/496 | 0/499
Other Adverse Events (participants affected / at risk) | 0/496 | 0/499

LIMITATIONS AND CAVEATS:
Low prevalence of HBV infection; individuals with barriers to healthcare were underrepresented; Quick Profile anti-HBsAb rapid test unable to confirm nonimmunized status; intervention had same-day blood draws, which is not done in routine practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No